CLINICAL TRIAL: NCT00546494
Title: A Study Of The Utility Of Effexor® (Venlafaxine) In Achieving Response And Maintaining Remission Among Taiwanese Patients With Depression
Brief Title: Study Evaluating Effexor® (Venlafaxine) in Achieving Response and Maintaining Remission
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0600B-101547
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Venlafaxine Hydrochloride

INTERVENTIONS:
Drug: Effexor® (Venlafaxine)

SUMMARY:
This is a study to determine the utility of Effexor® (venlafaxine) in achieving response, including time to response, maintaining remission, and time to remission as measured by the 17-item Hamilton Rating Scale for Depression (HAM-D) and to determine the utility of Effexor® (venlafxine) on the various cluster of symptom scales in the 17-item HAM-D.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients meeting criteria for a diagnosis of major depression, single or recurrent episode as described by the DSM-IV manual (appendix 1).
* A HAM-D 17 total score of at least 16 at baseline (DSM-IV manual, appendix 2).
* Patients above 18 years of age who meet the eligibility requirements.

EXCLUSION CRITERIA:

* Patients taking MAOI's within 2 weeks prior to the survey.
* Patients known to be suffering from bipolar disorder or schizophrenia.
* Patients who are treatment-resistant, i.e., in the past 3 years have failed (a) three previous adequate trials of greater than or equal to 2 classes of antidepressant medication, or (b) electroconvulsive therapy.
* Drug or alcohol dependence or abuse in the past 6 months per DSM IV criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350
Dates: Start 2004-02; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Primary efficacy variable will be the proportion of patients with remission defined as a HAM-D score of less than or equal to 7 at 8 weeks of treatment.

SECONDARY OUTCOMES:
Safety and tolerability will be assessed based on adverse events that occurred during the survey for all patients who received at least one dose of Effexor®.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer